CLINICAL TRIAL: NCT06652009
Title: Efficacy of Radical Radiotherapy Compared with Surgical Treatment in Patients with Upper Tract Urothelial Carcinoma: a Prospective Cohort Study
Brief Title: Radical Radiotherapy Versus Radical Surgery for UTUC
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LI xiaoying, Vice Director of the Department of Radiation Oncology, Peking University First Hospital
Other Study IDs: LUXUS6.0
Record Dates: First submitted 2024-09-12; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Renal Pelvis Cancer
Keywords: Renal pelvis carcinoma; Radical radiotherapy; Radical surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Radical surgery group: Patients undergo radical nephroureterectomy
  Interventions: Other: Radical nephroureterectomy
- Radical radiotherapy cohort: Patients undergo radical radiotherapy with stereotactic body radiation therapy (SBRT) or moderately segmented radiotherapy
  Interventions: Radiation: Radical radiotherapy

INTERVENTIONS:
Other: Radical nephroureterectomy — Radical nephroureterectomy
  Groups: Radical surgery group
Radiation: Radical radiotherapy — Radical radiotherapy with stereotactic body radiation therapy (SBRT) or moderately segmented radiotherapy
  Groups: Radical radiotherapy cohort

SUMMARY:
This study is a prospective cohort study, and the proposed plan is to recruit 30 patients with radical radiotherapy for renal pelvic ureteral cancer, according to the actual clinical situation, enrolling the same period of time to choose the operation of the elderly, combined with the risk of anaesthesia or regional lymph node metastasis of the patients, initially tentatively set at 60. The patients were divided into the surgery group and radiotherapy group according to the actual choice of treatment. In the control group, standard nephroureterectomy was used, and in the experimental group, stereotactic body radiation therapy (SBRT) or moderately segmented radical radiotherapy was used.

DETAILED DESCRIPTION:
1) No lymph node metastasis Choose SBRT radiotherapy as much as possible Tumour PTV 50Gy/10f; if the tumour is close to the intestine, the radiotherapy dose can be appropriately reduced 40-50Gy/8-10f; to ensure intestinal safety 2）With regional lymph node metastasis Renal pelvis tumour: tumour PGTV 62.5Gy/25f; for tumour larger than 3cm P-SBRT radiotherapy is feasible, SBRT 18-24Gy/3-4f; Affected kidney + para-abdominal aorta + common iliac lymph node drainage area 47.5Gy/25f; metastatic lymph nodes 62.5Gy/25f.

3) Routinely segmented normal tissue limits are as follows: Contralateral kidney V20<15% Dmean 15Gy Duodenum Dmax<50Gy Jejunum/ileum/colon V50<5% Dmax<52Gy Spinal cord Damx <40Gy Liver At least 700cc volume should receive a dose <25Gy

SBRT segmentation Normal tissue limits are as follows:

Duodenum Dmax<32Gy; V18<5cc Jejunum/ileum/colon Dmax<35Gy; V19.5<5cc Stomach Dmax<32Gy; V18<5cc (4) Short-term efficacy judgement: 1 month after radiotherapy to review imaging, short-term efficacy based on RECIST1.1 criteria, partial remission (PR partial regression) or complete remission (CR complete regression); disease-free survival is defined as the period after treatment to the emergence of recurrence in the radiotherapy field, intra-urethral recurrence (except bladder recurrence) or Regional lymph node metastases at first recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Uroepithelial carcinoma of the renal pelvis or ureter supported by clinical symptoms, imaging, histopathology, urocytology, or fluorescence in situ hybridisation (FISH), or those who satisfy FISH positivity despite the absence of pathology or the patient's refusal to be punctured and who are judged to have a renal pelvic or ureteral carcinoma by an imaging physician and a urologist on the basis of CTU or MRU or PETCT; No distant metastases were detected on full screening; Patients who are unable to undergo surgical treatment due to poor general condition, inability to be anaesthetised or to tolerate surgery, or refusal to undergo surgery; patients who are over 70 years old; or patients who are less than 70 years old combined with underlying diseases or the presence of regional lymph node metastasis, etc. who are otherwise unable to undergo radical surgery; Expected survival ≥ 6 months; Willingness and ability to comply with trial and follow-up procedural arrangements; voluntarily agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Previous abdominopelvic radiotherapy; Other serious, uncontrolled concomitant disease that may affect adherence to the protocol or interfere with interpretation of results; Other malignancies within 5 years prior to the start of study dosing, with the exception of malignancies that can be expected to resolve with treatment (including, but not limited to, adequately treated thyroid cancer, cervical cancer in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated by radical surgery); estimated that patients' adherence to participation in this clinical study was insufficient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ureteral cancer of the renal pelvis in patients with advanced age, combined anaesthetic risk or regional lymph node metastases
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative changes in renal function(eGFR) | Immediately postoperatively, 1 month and 6-12 months postoperatively
  Postoperative changes in renal function(eGFR)

SECONDARY OUTCOMES:
Adverse effects | 1 month after the start of treatment until the end of treatment
  Adverse effects related to radiotherapy and surgery
OS | Until the end of the project, an average of 5 years; a mid-term analysis is usually implemented at the 3rd year.
  Overall survival
PFS | Until the end of the project, an average of 5 years; a mid-term analysis is usually implemented at the 3rd year.
  Progression-free survival
Local response rate(LRR) | 1 month and 1 year after treatment
  Local response rate(LRR)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Departmeng of Urology, Peking University First Hospital, Beijing
  - Department of Radiotherapy Oncology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol